CLINICAL TRIAL: NCT00747864
Title: Relationship of Gestational Age and Urine Concentration of S100B in Preterm and Term Infants in the First Week of Life
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Joanna Beachy Ph.D., M.D., University of Utah
Other Study IDs: 14083
Record Dates: First submitted 2008-09-03; First posted 2008-09-05 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Preterm and Term Infants
Keywords: Gestational Age; Urine; Concentration; of S100B
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
S100B, a calcium-binding protein, is found predominantly in the central nervous system (CNS) and is increased in CSF and blood after CNS injury. There are two objectives to this study. 1) To complement our previous study, is urine S100B concentration correlated with gestational age in infants born at > 28 weeks gestation during the first week of life? 2) Is the urine concentration of S100B affected by intracranial pathology in this gestational age range? Elevation of urine concentration of S100B may be an indicator that the infant will develop serious intracranial pathology and may allow for early initiation of treatment to potentially decrease morbidity.

DETAILED DESCRIPTION:
S100B is a low molecular weight calcium binding protein found predominantly in the central nervous system (CNS), specifically astroglial cells.[1] S100B plays a role in calcium-dependent information processing and intracellulary is involved in the regulation of cytoskeleton and cell morphology.[1] S100B is secreted by astrocytes and exhibits dose dependent extracellular cytokine functions. In tissue culture at nanomolar concentration, S100B stimulates neuronal growth, development, and regeneration and protects against degeneration. At micromolar concentration, S100B is neurotoxic [2] and stimulates apoptosis potentially through interaction with RAGE receptor, by induction of NO synthase, and through the caspase cascade.

The evidence to support the S100B's role in development and maturation of the CNS is that S100B is differentially distributed in different cortical regions of the brain during fetal development and increases in concentration during gestation.[3] It is postulated that early in development, S100B stimulates glial cell proliferation while later it leads to extension of neurites, regulation of fiber sprouting, formation/maintenance of synapses, and maturation of glial cells.[1] Cord blood concentration of S100B has been shown to be inversely related to gestational age between 27 to 42 weeks gestation.[4] Thirty term infants (37-42 weeks) had mean cord blood S100B concentration of 0.47 ug/L (range 0-1.5ug/L) while 28 preterm infants (27-36 weeks) had a mean cord blood concentration of 1.14ug/L (range 0.5 and 2.7 ug/L). Higher serum concentration of S100B in preterm infants may be due the physiologic increase noted during development and/or lack of integrity of the blood-brain barrier.

S100B is released from damaged astroglial cells and may reflect neuronal damage.[5,6] Concentration of S100B is elevated in cerebrospinal fluid (CSF) of adult patients within 48 hours after infarction and remains elevated for at least 7 days after the event.[6] S100B is also elevated in CSF for the first 3 days after traumatic brain injury [7] and subarachnoid hemorrhage.[8] Due to its low molecular weight, S100B readily crosses a dysfunctional blood-brain barrier and serum concentration of S100B is significantly increased in adult patients after traumatic brain injury [9], stroke [10], or cardiac arrest.[5] Serum S100B rises for 2-4 days after brain trauma or infarct and its concentration correlates with size of damage as identified by CT scan. [9,10] After cardiac arrest, serum S100B concentration was statistically elevated by 30 minutes after initiation of CPR and continued to be significantly elevated in those patients who later exhibited brain damage by CT scan or neurological exam.[5] This significant elevation in serum S100B lasted for at least 7 days. In addition, serum S100B concentration correlated with morbidity [9] and neurological outcome.[10] While the t1/2 of S100B is ~2 hours in adults, persistently increased concentration of S100B in serum indicates continuous release from damaged cells.

The most common CNS trauma for preterm infants is intraventricular hemorrhage (IVH).[11] IVH originates in the microcirculation/capillary network of the germinal matrix. Altered cerebral blood flow secondary to poor cerebral autoregulation or systemic hypo- or hypertension, platelet and coagulation disturbances, infection, and decreased capillary integrity and vascular support have been implicated in the pathogenesis of IVH. IVH is graded (1-4) by extent of hemorrhage seen by ultrasound. In grade I IVH, the blood is confined to the germinal matrix. In Grade II IVH, blood is present in the germinal matrix and a small of blood is present in the ventricles. Grade III IVH occurs when the ventricles are filled with blood and dilated. In Grade IV IVH, blood extends into the brain parenchyma due to venous congestion of the terminal veins that border the lateral ventricles which leads to white matter necrosis. Grades I and II IVH are not associated with an increase in developmental abnormalities, but do not insure normalcy. Grades III and IV IVH (severe IVH) are highly associated with developmental delay, specifically spastic hemiplegia affecting the lower extremities more than the upper extremities due to the proximity of the hemorrhage to the descending motor fibers, and may also affect intellect. IVH, both mild (grade 1-2) and severe (grade 3-4) are rarely seen in infants with gestational age > 28 weeks due to the developmental involution of vessels in the germinal matrix which is the source of this hemorrhage.[11]

Due to its low molecular weight (10.5 kD) and high degree of solubility, S100B is excreted through the kidneys. It has been detected in the first void urine of infants between 26-42 weeks gestation with the most preterm infant exhibiting the highest concentration of S100B (3.17 ug/L).[12] Mean urine S100B concentration in term infants (n=60) was 0.07 ug/L. This study is confounded by no mention of intracranial pathology, insufficient number of preterm infants, and actual data was not shown. In another study, S100B was elevated in urine in preterm infants (29-35 weeks gestation) with IVH (grade 2-4) at birth and continued to increase over the subsequent 3 days when compared to control preterm infants.[13] The severity of IVH significantly correlated with the concentration of S100B in the urine. The highest level of S100B was seen in the five infants who died. An important limitation of the above cited study is insufficient patient enrollment to allow for correlation of both gestational age and presence of severe IVH on urine S100B concentration. Recently, we have shown that urine concentration of S100B is not elevated in very preterm infants (23-28 weeks gestation) without intracranial pathology.[pas abstract] However, very preterm infants with severe IVH (grade 3-4) had significantly elevated urine concentration of S100B on day 1.[14]

The specific aims of this study are to establish baseline S100B concentration in the urine of infants with gestational age > 28 weeks. In addition, the impact of intracranial pathology, that is IVH in preterm infants, will be further investigated. In the previous study, infants who developed necrotizing enterocolitis (NEC) had extremely high levels of S100B in the first week of life. NEC affects preterm infants, mostly 26-32 weeks gestation, and can result in death or markedly increased complications and prolonged length of stay. Secondary analysis of infants in this study will investigate if the development of NEC is significantly associated with a high concentration S100B in the urine. If this is true, one theory to explain this finding is that infants who develop NEC had an event around the time of birth that caused decrease intestinal perfusion allowing increased susceptibility to development of NEC.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at >28 weeks gestation will be eligible for enrollment in this study.

Exclusion Criteria:

* Infants with fetal malformations, chromosomal anomalies, clinically significant sepsis (retractable hypotension, neutropenia, and thrombocytopenia), or no urine output for the first 48 hours will be excluded.

Max Age: 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants born at >28 weeks gestation will be eligible for enrollment in this study. Infants with fetal malformations, chromosomal anomalies, clinically significant sepsis (retractable hypotension, neutropenia, and thrombocytopenia), or no urine output for the first 48 hours will be excluded. Infants that meet criteria will be enrolled in this study if the parent(s) sign the consent form. There are no patient safety or adverse event issues as this study is non-invasive and observational only.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2006-04; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Beachy, M.D., Principal Investigator — University of Utah